CLINICAL TRIAL: NCT05878925
Title: Nasal Olfactory Stimulation and Its Effect on Respiratory Drive in Preterm Infants - A Randomized Cross-over Study
Brief Title: Nasal Olfactory Stimulation and Its Effect on Respiratory Drive in Preterm Infants
Acronym: NOSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Bangerter-Rhyner Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NOSE
Record Dates: First submitted 2023-05-01; First posted 2023-05-30 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Apnea of Prematurity; Prematurity; Infant, Premature, Diseases
Keywords: Olfactory stimulation
MeSH Terms: conditions — Apnea; Premature Birth; Infant, Premature, Diseases | interventions — Odorants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To blind the study team and the medical team, identically looking pens will be provided with and without vanilla or strawberry aroma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aroma (Experimental): Preterm infants on CPAP support will be exposed to either vanilla or strawberry aroma. A pen with and without vanilla or strawberry aroma will be used to apply the aroma to the inner surface of the CPAP mask.
  Interventions: Other: Aroma
- Control (Placebo Comparator): Preterm infants on CPAP support will be exposed to placebo. The placebo pen will contain the carrier solution and natural coloring agents but no aroma.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Aroma — The study intervention is an olfactory stimulation with vanilla or strawberry aroma. The aroma will be applied to the inner surface of the nCPAP mask of preterm infants using designated scent pens every 3-4 hours over a period of 12 hours. The two aromas will be applied in blocks of 5 consecutive infants (5 infants vanilla, 5 infants strawberry, and so forth).
  Arms: Aroma
Other: Placebo — During the control intervention, identically looking placebo pens will be used to apply a colored carrier solution (without aroma) to the inner surface of the nCPAP mask of preterm infants in the same manner.
  Arms: Control

SUMMARY:
This trial analyzes the effect of an olfactory stimulation with vanilla or strawberry aroma compared to placebo on desaturations and bradycardia in preterm infants with apnea of prematurity. Infants on continuous positive airway pressure (CPAP) support will be included and the aroma will be applied to the inner surface of the CPAP mask using designated scent pens. The trial uses a cross-over design. Infants are randomised to begin the study with either aroma or placebo which will be applied into the breathing mask every 3 to 4 hours during 12 hours for each of the two intervention periods. Identically looking pens with either aroma or placebo are used and patients, parents, medical staff and the study team are blinded to this allocation. Infants are monitored with an oximetry sensor to measure peripheral oxygen saturation (SpO2) and pulse rate.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at birth: 23 0/7 to 31 6/7 weeks
* Postnatal age: >72 hours old
* Respiratory support: nCPAP
* Treatment with caffeine citrate for apnea of prematurity
* Written informed consent by one of the patient's parents

Exclusion Criteria:

* Olfactory impairment such as choanal atresia
* Intraparenchymal intracranial hemorrhage or intraventricular hemorrhage with ventricular dilation
* Culture-proven sepsis during the study period or any acute clinical deterioration requiring an intervention such as intubation or a new start of antibiotic treatment.
* Severe congenital malformation adversely affecting life expectancy

Min Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Paired difference in the combined number of desaturations and bradycardia | 12-hour recording periods for each intervention
  A desaturation is defined as a fall in the SpO2 to <80% for more than 10 seconds, a bradycardia is defined as a fall in heart rate <80 bpm for more than 10 seconds. Desaturation episodes and bradycardia separated by a time interval of five seconds or less will be counted as a single event. A desaturation episode as part of a bradycardia (or vice versa) will be counted as a two events. Peripheral oxygen saturation and heart rate will be monitored with an oximeter sensor placed around the infants' wrist or ankle and connected to the oximeter in 2 seconds averaging mode and maximum sensitivity.

SECONDARY OUTCOMES:
Paired difference in fraction of inspired oxygen (FiO2) | 12-hour recording periods for each intervention
  Paired difference in oxygen requirement between the two intervention periods. The FiO2 will be measured by the infant ventilator and documented in the patient data management system
Paired difference in mean peripheral oxygen saturation | 12-hour recording periods for each intervention
  Paired difference in oxygen saturation between the two intervention periods. Peripheral oxygen saturation and heart rate will be monitored with an oximeter sensor placed around the infants' wrist or ankle and connected to the oximeter in 2 seconds averaging mode and maximum sensitivity.
Paired difference in time spent with peripheral oxygen saturations <80% | 12-hour recording periods for each intervention
  Paired difference in total time spent with an oxygen saturation <80% between intervention periods. Peripheral oxygen saturation and heart rate will be monitored with an oximeter sensor placed around the infants' wrist or ankle and connected to the oximeter in 2 seconds averaging mode and maximum sensitivity.
Paired difference in time spent with heart rate <80 bpm | 12-hour recording periods for each intervention
  Paired difference in total time spent with a heart rate <80 beats per minute between intervention periods. Peripheral oxygen saturation and heart rate will be monitored with an oximeter sensor placed around the infants' wrist or ankle and connected to the oximeter in 2 seconds averaging mode and maximum sensitivity.
Paired difference in mean respiratory rate (as counted by nurses and manually) documented according to clinical routine) and heart rate | 12-hour recording periods for each intervention
  Paired difference in mean respiratory rate between intervention periods. Respiratory rate will be counted and documented by nurses every 4 to 8 hours according to clinical standard and documented in the patient data management system.
Paired difference in the apnea score documented by nurses | 12-hour recording periods for each intervention
  Paired difference in the apnea score (objective scoring system for the number and severity of apneas during a dedicated time frame) between intervention periods. Definition of the apnea score: Cumulative number of bradycardia <80 bpm and desaturations <80% during sleep and unimpaired wakefulness. Score 1 for event without need for intervention, score 2 for event requiring tactile stimulation, score 3 for event requiring increase of FiO2, score 8 for event requiring mask ventilation.
Paired difference in desaturations requiring stimulation or increase in FiO2 | 12-hour recording periods for each intervention
  Paired difference in the total number of desaturations requiring manual stimulation or an increase in supplemental oxygen between intervention periods. Manual stimulation will be documented by nurses in the patient data management system.
Paired difference in tolerance of enteral nutrition as assessed by gastric residuals (the amount of stomach liquid detected prior to the next meal, in mL) | 12-hour recording periods for each intervention
  Paired difference in amount of gastric residuals (mL) between intervention periods. Before each feed, nurses routinely aspirate orogastric tubes to check for the liquid volume and document the amount in mL in the patient data management system.

OTHER OUTCOMES:
Prespecified subgroup analyses of the primary outcome will be performed according to the type of aroma (vanilla or strawberry) that was administered. | 12-hour recording periods for each intervention
  A prespecified subgroup analysis for the primary outcome will be performed between infants receiving vanilla and strawberry aroma.

CONTACTS AND LOCATIONS:
Overall Officials: Janine Thomann, MD, Principal Investigator — Department of Neonatology, University Hospital and University of Zurich, Zurich, Switzerland
Locations (1):
- Department of Neonatology, Newborn Research, University Hospital and University of Zurich,, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No